CLINICAL TRIAL: NCT06551714
Title: The Effect of Neurophysiological Facilitation Techniques on Pulmonary Function, Respiratory Muscle Strength and Functional Capacity in The Early Stage After Open Heart Surgery
Brief Title: The Effect of Neurophysiological Facilitation Techniques on Health Parameters in Early Stages After Open Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dogus Universitesi (Other)
Responsible Party: Principal Investigator, Feyza Merakli, lecturer, Dogus Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DogusU
Record Dates: First submitted 2024-02-19; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Open Heart Surgery; Cardiovascular Disease; Physiotherapy
Keywords: Neurophysiological facilitation technique; Cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Phase 1 cardiac rehabilitation
  Interventions: Procedure: Phase 1 cardiac rehabilitation
- Study Group (Active Comparator): Neurophysiological facilitation techniques in addition to phase 1 cardiac rehabilitation techniques
  Interventions: Procedure: Phase 1 cardiac rehabilitation; Procedure: Neurophysiological facilitation techniques

INTERVENTIONS:
Procedure: Phase 1 cardiac rehabilitation — Day 1:Patients were informed about the surgery, positioning and mobilization.Range of motion (ROM), respiratory control, diaphragmatic breathing, pursed lip breathing, thoracal expansion exercises, assisted coughing,forced expiration techniques, which are the components of active breathing techniques cycle (ABTC), were taught.The use of incentive spirometry (IS) was demonstrated.Patients were performed 10 repetitions of IS exercises, and 5 repetitions ABTC and were asked to repeat them every hour.The patient was made to sit for 10 minutes and was walked 60 meters twice a day.
  2:ROM, IS and diaphragmatic breathing exercises were applied 10 times each.ABTC was repeated in 5 sets. 120 meters was walked 5 times during the day.
  3:Sitting time was increased to 30 minutes and walking distance was increased to 240 meters.5 steps were climbed.
  4:Walking distance was increased to 360 meters.One flight of stairs was climbed.Discharge training was given.
Procedure: Neurophysiological facilitation techniques — In addition to the phase 1 cardiac rehabilitation program for the group receiving neurophysiological facilitation (NPF) techniques:
  NPF techniques such as perioral stimulation, intercostal tension, anterior basal lift, vertebral pressure, moderate manual pressure and abdominal co-contraction were applied for ten times for ten seconds.
  Diaphragm facilitation exercise was performed by inhaling against resistance and holding the breath against resistance for 5 seconds.
  Unilateral and bilateral upper extremity proprioceptive neuromuscular facilitation (PNF) movements combined with breathing were performed.
  NPF techniques were performed 10 times each day throughout the treatment, while other applications (diaphragm facilitation, combined breathing exercise with upper extremity PNF technique and respiratory facilitation) were performed 5 times on the first day and 10 times on the other three days.
  Arms: Study Group

SUMMARY:
In this study, researchers aimed to investigate effects of neurophysiological facilitation on functional capacity and respiratory parameters of patients who underwent open heart surgery.

Do neurophysiological facilitation techniques improve individuals' respiratory parameters more than phase 1 cardiac rehabilitation?

Do neurophysiological facilitation techniques improve individuals' functional capacity more than phase 1 cardiac rehabilitation?

Researchers will apply phase 1 cardiac rehabilitation to both groups to see the effectiveness of neurophysiological facilitation techniques.

DETAILED DESCRIPTION:
In this study, researchers aimed to investigate effects of neurophysiological facilitation on functional capacity and respiratory parameters of patients who underwent open heart surgery.

The study was performed on 32 patients who underwent open heart surgery. Patients divided into two groups which study group (n=18) and control group (n=14).

Range of motion, breathing and mobilization exercises within the scope of phase 1 cardiac rehabilitation program were applied to the control group; in addition to the phase 1 cardiac rehabilitation program, neurophysiological facilitation techniques (perioral stimulation, intercostal tension, anterior basal lift, vertebral pressure, moderate manual pressure and abdominal co-contraction) were applied to the study group.

Sociodemographic features and disease-specific findings were recorded on the first postoperative day .

Vital signs, functional capacity, pulmonary function, fatigue and dyspnea of every patient were recorded before and after each treatment on the first four postoperative days.

Functional capacity was evaluated using Timed Up and Go (TUG) test and 2-Minutes Walking test (2MWT). Pulmonary function was examined using a peak flow meter and respiratory muscle strength was measured using an intraoral pressure measurement device. In addition, fatigue and dyspnea perception was measured using Modified Borg Scale.

Before the first day treatment and after the last day treatment of the four-day treatment, patients' fatigue severity were assessed with using Fatigue Severity Scale (FSS), anxiety and depression level with using Hospital Anxiety Depression Scale (HADS), fear of movement with using TAMPA Kinesiophobia Scale and life quality with using the Minnesota Heart Failure Questionnaire.

Before each treatment chest circumference measurements were taken, and the perceived pain severity was recorded using Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Having open heart surgery for the first time,
* Being between the ages of 18-75,
* Being fully cooperative

Exclusion Criteria:

* Having facial, sternum and rib fractures,
* Having chronic renal failure,
* Development of cerebrovascular accident,
* Having cognitive dysfunction,
* Development of deep vein thrombosis in the post-operative period,
* Having neuromuscular disease,
* Having an orthopedic disability,
* Intubation time longer than 24 hours,
* Staying in intensive care for more than 48 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
İnspiratory muscle strength | Before and after treatment on each day of treatment, up to 3 month
  Maximum Inspiratory Pressure (MIP) - pressure
Expiratory muscle strength | After and before treatment on each day of treatment, up to 3 month
  Maximum Expiratory Pressure (MEP) - pressure
2 Minute Walk Test | Before treatment on the first day of treatment and after treatment on the last day of treatment, up to 3 month
  It is walking as fast as the person can for 2 minutes without any assistance, at a safe distance of 30 meters. - meter
Time Up and Go (TUG) | first day of treatment before treatment and last day of treatment after treatment, up to 3 month
  The person gets up from the chair, walks 3 meters, comes back and sits on the chair. - minute
Vital sign | Before and after treatment on each day of treatment, up to 3 month
  Oxygen saturation
Respiratory frequency | Before and after treatment on each day, up to 3 month
  Number of times a person inhales and exhales in 1 minute. - number
Blood pressure | Before and after treatment on day of treatment, up to 3 month
  Blood pressure is the pressure of blood within the arteries of the circulatory system. - pressure
Heart rate | Before and after treatment on each day of treatment, up to 3 month
  Number of times a person heart rate in 1 minute. - number
Life quality | Before treatment on the first day of treatment and after treatment on the last day of treatment, up to 3 month
  The Minnesota Living with Heart Failure Questionnaire
Depression | Before treatment on the first day of treatment and after treatment on last day of treatment, up to 3 month
  Beck's depression inventory
Symptom | Before and after treatment on each day of treatment, up to 3 month
  Dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Cirak, Prof. Dr., Principal Investigator — Istinye University; Feyza merakli, Study Director — Istinye University
Locations (1):
- Lokman Hekim Akay Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, Informed Consent Form, Statistical Analysis Plan and Clinical Study Report will be shared upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will remain open for 1 year.
Access Criteria: To be a journal in Science Citation Index (SCI), Emerging Sources Citation Index (ESCI) categories